CLINICAL TRIAL: NCT02871336
Title: Pancreatic Surgical Database
Acronym: CHIRPAN
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: CHIRPAN
Record Dates: First submitted 2016-08-03; First posted 2016-08-18 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Pancreatic Neoplasms
Keywords: Cata collection; Pancreatic cancer surgery
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Data collection

SUMMARY:
This data base has been set in order to gather medical and surgical information from patients who have undergone surgery for pancreatic cancer, at Institut Paoli Calmettes or Assistance Publique des Hôpitaux de Marseille, France.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 ans
* Surgery for a pancreatic cancer

Exclusion Criteria:

* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a pancreatic cancer who has undergone surgery
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2014-11; Primary Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Optimization of the surgical care of the patients | 5 years
  Collection of clinical and surgical data for future research studies

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Turrini, MD,PhD, Principal Investigator — Institut Paoli-Calmettes; Vincent Moutardier, Principal Investigator — Assistance Publique des Hôpitaux de Marseille; Jean HARDWIGSEN, Principal Investigator — Assistance Publique des Hôpitaux de Marseille; Mehdi Ouassi, Principal Investigator — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches du Rhone, France

REFERENCES:
- [Derived] De Crignis L, Garnier J, Ewald J, Palen A, Piana G, Izaaryene J, Delpero JR, Turrini O. Preoperative liver arterial conditioning in patients scheduled for a Mayo Clinic class Ia distal pancreatectomy: embolization or ligation? HPB (Oxford). 2023 Apr;25(4):439-445. doi: 10.1016/j.hpb.2023.01.007. Epub 2023 Jan 20. PMID 36801197
- [Derived] Palen A, Garnier J, Ewald J, Delpero JR, Turrini O. Readmission after pancreaticoduodenectomy: Birmingham score validation. HPB (Oxford). 2023 Feb;25(2):172-178. doi: 10.1016/j.hpb.2022.08.002. Epub 2022 Aug 20. PMID 36437219